CLINICAL TRIAL: NCT02260804
Title: A Phase 3, Randomised, Parallel-group, Active-controlled, Double-blind Study to Compare Efficacy and Safety Between CT-P10 and Rituxan in Patients With Low Tumour Burden Follicular Lymphoma
Brief Title: To Compare Efficacy and Safety Between CT-P10 and Rituxan in Patients With Low Tumour Burden Follicular Lymphoma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-P10 3.4
Record Dates: First submitted 2014-10-05; First posted 2014-10-09 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-02

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — CT-P10; Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-P10 (Experimental): CT-P10, intervention 375mg/m2, intravenous, 4 cycles in induction period and additional 12 cycles in maintenance period
  Interventions: Biological: CT-P10
- Rituxan (Active Comparator): Rituxan, 375mg/m2 intravenous, 4 cycles in induction period, Rituxan for the first 6 cycles and CT-P10 for the last 6 cycles in maintenance period.
  Interventions: Biological: Rituxan

INTERVENTIONS:
Biological: CT-P10 — 375mg/m2, IV on day1 of 4 cycles in induction period, and 12 cycles in maintenance period.
  Arms: CT-P10
Biological: Rituxan — 375mg/m2, IV on day1 of 4 cycles in induction period, Rituxan for the first 6 cycles and CT-P10 for the last 6 cycles in maintenance period.
  Arms: Rituxan

SUMMARY:
To demonstrate that CT-P10 is similar to Rituxan in terms of efficacy as determined by overall response rate at 7 months

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of low tumour burden, CD20+ follicular lymphoma
* Ann Arbor Stage II, III or IV

Exclusion Criteria:

* Has receive rituximab
* Allergies or hypersensitivity to murine, chimeric, human or humanised proteins
* Previous treatment for NHL
* Any malignancy
* Current or recent treatment with any other investigational medicinal product or device
* pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2015-11-09 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2019-09-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SungHyun Kim, Study Director — Celltrion
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kwak LW, Sancho JM, Cho SG, Nakazawa H, Suzumiya J, Tumyan G, Kim JS, Menne T, Mariz J, Ilyin N, Jurczak W, Lopez Martinez A, Samoilova O, Zhavrid E, Yanez Ruiz E, Trneny M, Popplewell L, Ogura M, Kim WS, Lee SJ, Kim SH, Ahn KY, Buske C. Efficacy and Safety of CT-P10 Versus Rituximab in Untreated Low-Tumor-Burden Follicular Lymphoma: Final Results of a Randomized Phase III Study. Clin Lymphoma Myeloma Leuk. 2022 Feb;22(2):89-97. doi: 10.1016/j.clml.2021.08.005. Epub 2021 Aug 28. PMID 34686445
- [Derived] Ogura M, Sancho JM, Cho SG, Nakazawa H, Suzumiya J, Tumyan G, Kim JS, Lennard A, Mariz J, Ilyin N, Jurczak W, Lopez Martinez A, Samoilova O, Zhavrid E, Yanez Ruiz E, Trneny M, Popplewell L, Coiffier B, Buske C, Kim WS, Lee SJ, Lee SY, Bae YJ, Kwak LW. Efficacy, pharmacokinetics, and safety of the biosimilar CT-P10 in comparison with rituximab in patients with previously untreated low-tumour-burden follicular lymphoma: a randomised, double-blind, parallel-group, phase 3 trial. Lancet Haematol. 2018 Nov;5(11):e543-e553. doi: 10.1016/S2352-3026(18)30157-1. PMID 30389036
- See also: Related Info — http://www.celltrion.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 402 participants were screened for the study. Of those, 144 participants failed screening and 258 participants were enrolled in the study.
Groups:
- CT-P10: CT-P10 375mg/m2, IV, 4 cycles in induction period and additional 12 cycles in maintenance period
- Rituxan: Rituxan, 375mg/m2, IV, 4 cycles in induction period, Rituxan for the first 6 cycles and CT-P10 for the last 6 cycles in maintenance period.
Period: Induction Study Period
Arm/Group | CT-P10 | Rituxan
Started | 130 | 128
Completed | 128 | 128
Not Completed | 2 | 0
Not completed — Protocol Violation | 2 | 0
Period: 1st Year of the Maintenance Period (MP1)
Arm/Group | CT-P10 | Rituxan
Started | 123 (Five subjects completed the induction period but did not initiate this period in the CT-P10 group.) | 120 (Eight subjects completed the induction period but did not initiate this period in the Rituxan group.)
Completed | 111 | 105
Not Completed | 12 | 15
Not completed — Lack of Efficacy | 6 | 9
Not completed — Adverse Event | 3 | 1
Not completed — Physician Decision | 1 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Period: 2nd Year of the Maintenance Period (MP2)
Arm/Group | CT-P10 | Rituxan
Started | 110 (One subject completed the MP1 but did not initiate this period in the CT-P10 group.) | 103 (Two subjects completed the MP1 but did not initiate this period in the Rituxan group.)
Completed | 101 | 97
Not Completed | 9 | 6
Not completed — Lack of Efficacy | 6 | 5
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CT-P10 | Rituxan | Total
Number analyzed (Participants) | 130 | 128 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (12.68) | 57.7 (11.53) | 57.7 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 71 | 135
  Male | 66 | 57 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 10 | 22
  Not Hispanic or Latino | 110 | 116 | 226
  Unknown or Not Reported | 8 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Primary Efficacy Endpoint - Overall Response Rate by 7 Months
Description: ORR was defined as the proportion of patients with the best response of complete response (CR), unconfirmed CR (CRu), or partial response (PR) by central review.
  Per 1999 IWG criteria, the disease status was assessed by using contrasted CT and/or MRI, and CR, CRu, and PR were defined as followings; CR=Disappearance of all clinical/radiographic evidence of disease: regression of lymph nodes to normal size, absence of B-symptoms, bone marrow involvement, and organomegaly, and normal LDH level; CRu=Regression of measurable disease: >75% decrease in SPD of target lesions and in each target lesions. no increase in the size of non-target lesions, neither new lesion nor organomegaly measured; PR=Regression of measurable disease: ≥50% decrease in SPD of target lesions and no evidence of disease progression.
Time Frame: During the Month 7 (up to Maintenance Cycle 3; Week 28)
Population: The ITT population consisted of all patients enrolled and randomly assigned to receive a study drug, regardless of whether or not any study drug dosing was completed.
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 130 | 128
Participants | 108 | 104
Statistical Analysis 1: Comparison: CT-P10; Test type: Equivalence — The equivalence margin of ±17% was predefined; Difference in proportion = 1.8, 90% CI 2-sided [-6.43 to 10.2]

2. Secondary Outcome: Secondary Efficacy Endpoint - ORR Over the Study Period
Description: ORR was defined as the proportion of patients with the best response of complete response (CR), unconfirmed CR (CRu), or partial response (PR).
  Per 1999 IWG criteria, the disease status was assessed by using contrasted CT and/or MRI, and CR, CRu, and PR were defined as followings; CR=Disappearance of all clinical/radiographic evidence of disease: regression of lymph nodes to normal size, absence of B-symptoms, bone marrow involvement, and organomegaly, and normal LDH level; CRu=Regression of measurable disease: >75% decrease in SPD of target lesions and in each target lesions. no increase in the size of non-target lesions, neither new lesion nor organomegaly measured; PR=Regression of measurable disease: ≥50% decrease in SPD of target lesions and no evidence of disease progression.
Time Frame: up to 27 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 130 | 128
Participants | 109 | 112

3. Secondary Outcome: Secondary PD Endpoint - B-cell Kinetics (B-cell Depletion and Recovery)
Description: B-cell kinetics were demonstrated by median values of B-cell counts. Any values below the LLoQ were set as LLoQ which was 20 cells/μL.
Time Frame: Baseline, Induction Cycle 1 (predose, 1 hr postdose), Induction Cycle 2 to 4 (predose), EOT1/EOT2 (anytime), Maintenance Cycle 1 to 2 (predose, 1hr postdose) and Maintenance Cycle 3 (predose).
Population: The PD population consisted of all patients who received at least 1 dose (full) of study drug and had at least 1 posttreatment PD result.
Measure: Median (Inter-Quartile Range); unit: cells/uL
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 128 | 128
cells/uL
  Baseline: number analyzed (Participants) | 120 | 123
  Baseline | 95.0 [56.0 to 171.5] | 120.0 [64.0 to 182.0]
  Induction Cycle 1 (1hr after end of infusion): number analyzed (Participants) | 114 | 111
  Induction Cycle 1 (1hr after end of infusion) | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Induction Cycle 2 (predose): number analyzed (Participants) | 122 | 121
  Induction Cycle 2 (predose) | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Induction Cycle 3 (predose): number analyzed (Participants) | 122 | 124
  Induction Cycle 3 (predose) | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Induction Cycle 4 (predose): number analyzed (Participants) | 121 | 122
  Induction Cycle 4 (predose) | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  EOT1 (anytime): number analyzed (Participants) | 126 | 125
  EOT1 (anytime) | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Maintenance Cycle 1 (predose): number analyzed (Participants) | 113 | 121
  Maintenance Cycle 1 (predose) | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Maintenance Cycle 1 (1hr after end of infusion): number analyzed (Participants) | 105 | 108
  Maintenance Cycle 1 (1hr after end of infusion) | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Maintenance Cycle 2 (predose): number analyzed (Participants) | 112 | 113
  Maintenance Cycle 2 (predose) | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Maintenance Cycle 2 (1hr after end of infusion): number analyzed (Participants) | 107 | 108
  Maintenance Cycle 2 (1hr after end of infusion) | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]
  Maintenance Cycle 3 (predose): number analyzed (Participants) | 112 | 109
  Maintenance Cycle 3 (predose) | 20.0 [20.0 to 20.0] | 20.0 [20.0 to 20.0]

4. Secondary Outcome: Secondary PK Endpoints - Cmax
Time Frame: 1, 2, 3, 4, 12, 20 weeks (predose, 1 hr post dose), EOT1/EOT2 (anytime during the day) and 28 week (predose)
Population: The PK population consisted of all patients who received at least 1 dose (full) of study drug and had at least 1 posttreatment PK result.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 128 | 128
μg/mL
  Induction Cycle 1 | 212.86 (50.64) | 217.38 (56.33)
  Induction Cycle 2: number analyzed (Participants) | 127 | 127
  Induction Cycle 2 | 283.35 (53.84) | 285.98 (62.26)
  Induction Cycle 3: number analyzed (Participants) | 125 | 126
  Induction Cycle 3 | 327.32 (71.05) | 341.59 (77.95)
  Induction Cycle 4: number analyzed (Participants) | 125 | 128
  Induction Cycle 4 | 373.46 (70.50) | 383.05 (83.86)
  Maintenance Cycle 1: number analyzed (Participants) | 120 | 117
  Maintenance Cycle 1 | 256.97 (65.61) | 265.03 (53.73)
  Maintenance Cycle 2: number analyzed (Participants) | 119 | 116
  Maintenance Cycle 2 | 239.70 (65.72) | 249.86 (69.02)

5. Secondary Outcome: Secondary PK Endpoints - Ctrough
Time Frame: 1, 2, 3, 4, 12, 20 weeks (predose, 1 hr post dose), EOT1/EOT2 (anytime during the day) and 28 week (predose)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 128 | 128
μg/mL
  Induction Cycle 1: number analyzed (Participants) | 126 | 127
  Induction Cycle 1 | 64.66 (24.88) | 72.94 (40.39)
  Induction Cycle 2: number analyzed (Participants) | 127 | 126
  Induction Cycle 2 | 113.23 (34.60) | 120.92 (36.02)
  Induction Cycle 3: number analyzed (Participants) | 125 | 128
  Induction Cycle 3 | 149.53 (43.65) | 161.80 (43.91)
  Induction Cycle 4: number analyzed (Participants) | 122 | 125
  Induction Cycle 4 | 34.78 (33.58) | 31.38 (19.15)
  Maintenance Cycle 1: number analyzed (Participants) | 120 | 117
  Maintenance Cycle 1 | 22.68 (37.22) | 21.35 (20.90)
  Maintenance Cycle 2: number analyzed (Participants) | 118 | 110
  Maintenance Cycle 2 | 16.96 (9.61) | 18.37 (10.86)

6. Secondary Outcome: Secondary Efficacy Endpoint - Progression-free Survival (PFS)
Description: PFS was defined as the interval between randomization and disease progression/relapse by IWG 1999 (at least a 50% increase of any single nodal after smallest decrease) or death from any cause, whichever occurred first. Locally reviewed data was used for the secondary efficacy analyses.
Time Frame: Overall study period (Baseline, Month 3, 7, 13, 19 27, and every 6 months thereafter).
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 130 | 128
Proportion of Participants
  12 months | 0.93 [0.87 to 0.96] | 0.89 [0.82 to 0.93]
  24 months | 0.88 [0.81 to 0.92] | 0.83 [0.75 to 0.89]
  36 months | 0.80 [0.70 to 0.87] | 0.68 [0.54 to 0.79]

7. Secondary Outcome: Secondary Efficacy Endpoint - Overall Survival (OS)
Description: Overall survival was defined as the interval between randomization and death from any cause. Locally reviewed data was used for the secondary efficacy analyses.
Time Frame: Overall study period (median follow-up of 29.2 months)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 130 | 128
Proportion of Participants
  12 months | 0.98 [0.93 to 0.99] | 0.98 [0.94 to 1.00]
  24 months | 0.98 [0.93 to 0.99] | 0.98 [0.94 to 1.00]
  36 months | 0.98 [0.93 to 0.99] | 0.97 [0.89 to 0.99]
  42 months | 0.98 [0.93 to 0.99] | 0.97 [0.89 to 0.99]

8. Secondary Outcome: Secondary Efficacy Endpoint - Time-to Progression (TTP)
Description: Time to progression was defined as the interval between randomization and disease progression/relapse by IWG 1999 (at least a 50% increase of any single nodal after smallest decrease) or death as a result of lymphoma, whichever occurred first. Locally reviewed data was used for the secondary efficacy analyses.
Time Frame: Overall study period (Baseline, Month 3, 7, 13, 19 27, and every 6 months thereafter).
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | CT-P10 | Rituxan
Number analyzed (Participants) | 130 | 128
Proportion of Participants
  12 months | 0.94 [0.88 to 0.97] | 0.89 [0.83 to 0.94]
  24 months | 0.89 [0.82 to 0.94] | 0.84 [0.76 to 0.89]
  36 months | 0.82 [0.72 to 0.88] | 0.68 [0.54 to 0.79]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and Serious adverse events (SAEs) were to be collected from the date the ICF was signed until up to 30 days from the last dose of the study drug, regardless of the relationship to the study drug. data from the overall study period (median follow-up of 29.2 months) are presented.
Arm/Group | CT-P10 | Rituxan
All-Cause Mortality (participants affected / at risk) | 3/130 | 3/128
Serious Adverse Events (participants affected / at risk) | 14/130 | 14/128
Other Adverse Events (participants affected / at risk) | 93/130 | 86/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P10 (N=130) | Rituxan (N=128)
Angina unstable (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Peptic ulcer perforation (Gastrointestinal disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Genital prolapse (Reproductive system and breast disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Gastrointestinal surgery (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CT-P10 (N=130) | Rituxan (N=128)
Neutropenia (Blood and lymphatic system disorders) | 10 | 7
Abdominal pain (Gastrointestinal disorders) | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 9 | 11
Nausea (Gastrointestinal disorders) | 7 | 11
Fatigue (General disorders) | 10 | 13
Herpes virus infection (Infections and infestations) | 7 | 5
Influenza (Infections and infestations) | 3 | 8
Lower respiratory tract infection (Infections and infestations) | 6 | 11
Upper respiratory tract infection (Infections and infestations) | 31 | 29
Urinary tract infection (Infections and infestations) | 9 | 13
Infusion related reaction (Injury, poisoning and procedural complications) | 42 | 39
Alanine aminotransferase increased (Investigations) | 7 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Headache (Nervous system disorders) | 6 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Hypertension (Vascular disorders) | 10 | 6

LIMITATIONS AND CAVEATS:
In this study, TTE endpoints were secondary endpoints and were not powered. As medians of PFS, TTP, and OS were not reached in both treatment groups, longer follow-up is needed to ascertain the median time for TTE parameters of PFS, TTP, and OS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A confidentiality and non-disclosure agreement (CDA) was executed between Celltrion, Inc. and some PIs who have participated in publications funded by the sponsor for academic purposes for a period that is more than 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2017-06-28): https://cdn.clinicaltrials.gov/large-docs/04/NCT02260804/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-17): https://cdn.clinicaltrials.gov/large-docs/04/NCT02260804/SAP_001.pdf